CLINICAL TRIAL: NCT06185322
Title: The Effectiveness of Exercise on Neck Pain, Posture, Function and Quality of Life in Individuals With Upper Cross Syndrome: a Randomized Double Blind Control Study
Brief Title: Effectiveness of Exercise in the Treatment of Upper Cross Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Selin Ozen, Associate Professor Doctor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KA23/139
Record Dates: First submitted 2023-12-06; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Upper Cross Syndrome
Keywords: upper cross syndrome; forward head position; posture; neck pain; cervicalgia; pain ,cervical; posture balance
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus; Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The physiatrist who will initially assess, diagnose and collect outcome measures, will be blind to the study group of the patient.
  The patient will not know whether they are receiving the detailed exercise program or conventional exercise program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck strengthening exercises group (Active Comparator): 10 sessions of physical therapy over two weeks.Each session will consist of 20 minutes of hotpack and transcutaneous electrical nerve stimulation and 10minutes of therapeutic ultrasound. Exercise sessions lasting 20minutes will consist of conventional neck isometric strengthening exercises under the supervision of a single physiotherapist. These exercises will be repeated 5 times each, twice daily. A brochure depicting each exercise,accompanied by a description,will be given to the patient.The patient will continue with the exercise program for 3 months and be reminded once a week via telephone.
  Interventions: Other: Physical therapy program with conventional neck strengthening exercises
- Upper Cross Syndrome exercises group (Experimental): 10sessions of physical therapy over two weeks.Each session will consist of 20minutes of hotpack and transcutaneous electrical nerve stimulation and 10minutes of therapeutic ultrasound.Exercise sessions lasting 20minutes will consist of stretching and strengthening exercises under the supervision of a single physiotherapist.Strengthening exercises for the deep neck flexors,upper and middle trapezius,serratus anterior will be performed by the patient.Ten repetitions of each exercise,three times daily will be recommended.Stretching exercises will include those for the upper trapezius,pectoralis majör,levator scapula,suboccipital and sternocleidemastoid muscles and izometric neck flexion-extension exercises.These will be repeated 5times each,twice daily.A brochure depicting each exercise,accompanied by a description,will be given to the patient.The patient will continue with the exercise program for 3 months and be reminded once a week via telephone.
  Interventions: Other: Physical therapy program with upper cross syndrome specific exercises

INTERVENTIONS:
Other: Physical therapy program with upper cross syndrome specific exercises — Ten physical therapy sessions consisting of electrotherapy and upper cross syndrome -specific exercise program.
  Arms: Upper Cross Syndrome exercises group
Other: Physical therapy program with conventional neck strengthening exercises — Ten physical therapy sessions consisting of electrotherapy and conventional neck strenthening exercises
  Arms: Neck strengthening exercises group

SUMMARY:
Upper cross syndrome (UCS) is a common postural deformity characterized by a change in neck, torso and shoulder muscle activity and shoulder movement. UCS results in a shortening of the upper back and chest muscles as well as the muscles which provide movement to the shoulder blade. This is accompanied by weakness of the upper back muscles, shoulder blade stabilizor muscles and deep neck muscles. The resultant muscle imbalance leads to elevation of the shoulders, elongation of the neck and rounding of the back.

The change in posture which occurs in UCS changes the biomechanics of the neck and upper back and can results in neck pain, adverse effects on daily activities and productivity. To date, studies have been done on treatment of elongation of the neck using muscle relaxation techniques and manipulation of the local structures. To date, there is no study which investigates the efficacy of a specific exercise program targeting the muscles affected by UCS. The aim of this study is to investigate the effects of UCS-specific exercises on neck-back pain, cervical posture, disability and quality of life.

DETAILED DESCRIPTION:
Upper cross syndrome (UCS) is a common postural deformity characterised by a change in neck, torso and scapular muscle activity and scapular mobility. UCS results in a shortening of the upper trapezius, pectoralis majör and levator scapula muscles and weakness of the rhomboid, serratus anterior, middle and lower trapezii and deep cervical muscles such as the scalene muscles. The resultant muscle imbalance results in elevation and protraction of the shoulders, protraction of the neck and increase in kyphosis of the thoracic spine.

The change in posture seen in UCS reuslts in a change in the biomechanics of the vertebral bodies, neural arcus, musculature, faset joints, ligaments and discs which in turn can result in pain. Neck pain can negatively affect activities of daily living and function, causing disabiltiy and thus having a detrimental affect quality of life and productivity. Furthermore, studies have shown that UCS is frequently seen occuring in individuals with facet joint degeneration, myofacial pain syndrome and cervical radiculopathy. , In the literature, forward head position is treated craniocervical flexion training, muscle energy techniques, cervical coordination exercises, mobilization, manipulation and stabilization exercises. However, to date, there are no studies which investigate the effect of specific exercises aimed at resolving the muscle imblance which occurs in UCS. The aim of this study is to investigate the effects of UCS-specific exercises on neck-back pain, cervical posture and alignment, disability and quality of life. ,

ELIGIBILITY:
Inclusion Criteria: Male and female patients between the ages of 30-50 years attending the outpatient clinic of our physical medicine and rehabilitation department with neck and back pain with upper cross syndrome on examination.

Exclusion Criteria:

* History of cervical spine trauma or surgery
* Congenital postural deformity
* A history of inflammatory arthritis
* A diagnosis of torticollis, vertigo, pregnancy, vertebrobasilar insufficiency, heart failure, ischaemic heart disease, hypertension.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale measurement of severity of neck pain | Before physcial therapy treatment is commenced, after 10 sessions of physical therapy has been completed (2 weeks after commencement of therapy), three months after physical therapy has been completed.
  A subjective measure of neck pain severity in the past week measured using a visual analogue scale from 0-100mm. 0mm signifies no pain, 100mm signifies the worst pain imaginable.

SECONDARY OUTCOMES:
Neck disability index (NDI) | Before physcial therapy treatment is commenced, three months after physical therapy has been completed.
  A subjective measure of effect of neck pain on disability and activities of daily living. A ten part questionnaire on intensity of neck pain, effects of neck pain on self-care, heavy lifting, association between neck pain and headaches, ability to work and sleep. Each question scores between 0-5 with an increase in score signifying worsening disablity.
Nottingham Health Profile (NHP) | Before physcial therapy treatment is commenced, three months after physical therapy has been completed.
  A quality of life measure focusing on the effects of a health issue on daily activities. Measures of pain and energy levels, emotional wellbeing, sleep quality, social isolation and physical activity are conducted. A total score between 0-600 is obtained. Higher scores signify poorer quality of life. ,
Goniometric measurement of cervical range of motion | Before physcial therapy treatment is commenced, three months after physical therapy has been completed.
  Goniometric measurement of cervical flexion and extension
Occiput to wall distance and tragus to wall distance | Before physcial therapy treatment is commenced, three months after physical therapy has been completed.
  Measurement of the distance between the occiput and wall and tragus and wall in the sagittal plane when standing with feet against wall, head in the neutral position as a measure of cervical mobility and thoracic kyphosis.
Radiographic evaluation of cervical posture and cervicothoracic alignment: Measure of cervical lordotic angle | Before physcial therapy treatment is commenced, three months after physical therapy has been completed.
  Cervical lordotic angle will be evaluated by measuring the Cobb angle and absolute rotation angle (ARA). Cobb angle will be measured using a lateral cervical radiograph. A line will be drawn parallel to the C2 and C7 vertebral endplate. A second line will bisect these lines. The angle between the two bisecting lines is the Cobb angle. The ARA is formed by the intersection of tangents drawn at the posterior body margins of C2 and C7.
  To investigate the position of the head in the sagittal plane and sagittal alignment of the spine, the sagittal vertical axis (SVA) - distance between the posterior superior corner of C7 and a plumb line dropped from C2 - will be measured.
Radiographic evaluation of cervicothoracic alignment | Before physcial therapy treatment is commenced, three months after physical therapy has been completed.
  SCA refers to a new sagittal parameter, defined as the angle between a line from the sella turcica center and C7 endplate and the C7 plateau line.